CLINICAL TRIAL: NCT06582537
Title: Ex Vivo Genetic Correction of LAMA2 Mutation(s) in Myogenic Stem Cells of Patients with Merosin-deficient Congenital Muscle Dystrophy Type 1a (MDC1a)
Brief Title: LAMA2 Genetic Correction
Status: Completed | Type: Observational
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: MABS03
Record Dates: First submitted 2022-01-11; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-07

CONDITIONS: MDC1A
Keywords: MDC1A; LAMA2; Muscular Dystrophy; Mesoangioblasts
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adult carriers of the LAMA2 c.5562+5G>C mutation
  Interventions: Procedure: Participants sample collection
- Healthy controls
  Interventions: Procedure: Participants sample collection

INTERVENTIONS:
Procedure: Participants sample collection — A skeletal muscle biopsy and a venous blood sample will be collected. The skin biopsy will be obtained during the incision needed for the muscle biopsy.

SUMMARY:
Merosin-deficient congenital muscle dystrophy type 1a (MDC1a), or LAMA2 muscular dystrophy (LAMA2-MD) is a severe autosomal recessive form of muscular dystrophy that is caused by homozygous or compound heterozygous mutations in the laminin alpha 2 (LAMA-2) gene. Many different LAMA-2 mutations have been reported. In most cases, MDC1a is diagnosed within the first year of life, and is characterized by hypotonia, delayed motor development and white matter abnormalities. Currently, no efficient treatment is available for this patient group. Generally, MDC1a patients with mutations causing a premature stop codon are most severely affected (early onset LAMA2-MD) and patients with missense mutations are generally affected more mild affected and more late-onset (late onset LAMA2-MD). However, large variation in disease severity and clinical course is observed, even between individuals with the same mutation, e.g. the LAMA2 c.5562+5G>C mutation, which is frequently observed in Dutch MDC1a patients. This study aims to isolate and culture fibroblasts and myogenic stem cells called mesoangioblasts from the skin and muscle biopsies of adult LAMA2 mutation carriers to explore if genetic correction of LAMA2 mutations using CRISPR-Cas9 can be achieved and subsequently assess the effect in vitro, as a first step towards therapy development.

ELIGIBILITY:
Inclusion Criteria:

* LAMA2 mutation carriers:
* Age >18 years
* Heterozygous or homozygous LAMA2 c.5562+5G>C mutation
* Written informed consent

Controls:

* Written informed consent
* Age >18 years
* No muscular dystrophy or other disease known to affect muscle morphology or function

Exclusion Criteria:

* MDC1a patients and controls:
* No informed consent
* Use of anti-coagulants, anti-thrombotics and other medication influencing coagulation
* Have a weekly alcohol intake of ≥ 35 units (men) or ≥ 24 units (women)
* Current history of drug abuse
* A history of strokes
* Significant concurrent illness
* Ongoing participation in other clinical trials
* Major surgery within 4 weeks of the visit
* Pregnant or lactating women
* Patients unable and/or unwilling to comply with treatment and study instructions
* Any other factor that in the opinion of the investigator excludes the patient from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will only include patients/controls living in The Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Compare RNA transcription of corrected and not corrected DNA | 1 day
  qPCR
Assess effect LAMA2 mutations on muscle protein quantity (amount of LAMA2) | 1 day
  LAMA2 immunostaining
Assess effect LAMA2 mutations on muscle protein quality (localization of LAMA2) | 1 day
  LAMA2 immunostaining
Assess effect LAMA2 mutations on muscle protein quantity (LAMA2 overall levels) | 1 day
  LAMA2 western blot
Assess effect LAMA2 mutations on muscle protein quality (fibrosis) | 1 day
  LAMA2 HE staining

SECONDARY OUTCOMES:
Verification of the LAMA2 mutations or exclusion of LAMA2 mutations in controls | 1 day
  DNA analysis
Blood markers to assess level of muscle inflammation, damage and regeneration in MDC1a patients: CK | 1 day
  ELISA assay
Blood markers to assess level of muscle inflammation, damage and regeneration in MDC1a patients: TNFa | 1 day
  ELISA assay
Blood markers to assess level of muscle inflammation, damage and regeneration in MDC1a patients: IL-6 | 1 day
  ELISA assay
Blood markers to assess level of muscle inflammation, damage and regeneration in MDC1a patients: SDF1 | 1 day
  ELISA assay

CONTACTS AND LOCATIONS:
Locations (1):
- Academisch Ziekenhuis Maastricht, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No